CLINICAL TRIAL: NCT04129528
Title: Investigator- and Subject-blinded, Randomized, Placebo-controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy Trial of CFZ533 in Pediatric and Young Adult Subjects With New Onset Type 1 Diabetes (T1DM)
Brief Title: Study of Safety and Efficacy of CFZ533 in Type 1 Diabetes Pediatric and Young Adult Subjects
Acronym: CCFZ533X2207
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCFZ533X2207; 2018-004553-25 (EudraCT Number)
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — iscalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CFZ533 (Active Comparator): Randomized in a 2:1 ratio: 2 Active / 1 Placebo
  Interventions: Drug: CFZ533
- Placebo (Placebo Comparator): Similar in appearance to active study drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CFZ533 — First dose is administered via intravenous infusion, subsequent doses are administered subcutaneously.
  Other Names: Iscalimab
  Arms: CFZ533
Other: Placebo — Placebo for active drug
  Arms: Placebo

SUMMARY:
The study was a Phase 2, multicounty, multicenter, non-confirmatory, investigator- and subject masked, randomized, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of CFZ533 on preservation of residual pancreatic β-cell function in new onset T1DM in pediatric and young adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, and if needed assent from the child on the trial, must be obtained before any assessment is performed.
2. Males and females aged between 12 and 21 years (inclusive, and enrolled in stages) at screening.
3. Body weight range from 30 to 125 kg (inclusive).
4. Evidence of one or more type 1 diabetes autoantibody(ies) against: glutamic acid decarboxylase (anti-GAD), protein tyrosine, phosphatase-like protein (anti-IA-2); zinc transporter 8 (anti-ZnT8); islet cell (cytoplasmic) (anti-ICA) at screening or baseline in the central laboratory OR historical clinical record of one or more of the T1DM diabetes autoantibodies. As part of the historical record insulin autoantibodies (IAA) may have been used as part of the autoantibody panel but the blood sample must have been obtained prior to or within one week of starting exogenous insulin treatment.
5. Able to receive first dose of study drug within 56 days of diagnosis of T1DM (which may be extended to within 100 days of diagnosis in the event a screening assessment needs to be confirmed or vaccine administered).
6. Peak stimulated C-peptide levels ≥0.2 nmol/L (0.6 ng/mL) following standard liquid mixed meal tolerance test (MMTT), to be conducted when the subject is metabolically stable, at least 2 weeks from diagnosis and within 56 days prior to randomization (or within 100 days of diagnosis in the event a screening assessment needs to be confirmed or vaccine is required).
7. Study participants are to complete all recommended immunizations with live, attenuated vaccine at least eight weeks prior and killed, inactivated vaccine at least two weeks prior to first dose with study drug and in accordance with local immunization guidelines. In the event a subject has not had all vaccinations recommended according to local guidance, the screening period may be extended beyond 56 days to allow these vaccinations to be administered, but first dose of study drug must be administered within 100 days of diagnosis of T1DM.
8. Must be willing to comply with the standard of care for diabetes management.
9. A negative pregnancy test at screening is required for all sexually mature female subjects prior to participation in the study.
10. Subject and/or guardian must be able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Diabetes forms other than auto immune type 1 such as maturity-onset diabetes of the young (MODY), latent autoimmune diabetes of the adult (LADA), acquired diabetes (secondary to medications or surgery), type 2 diabetes by judgement of the investigator.
2. Diabetic ketoacidosis within 2 weeks of the baseline MMTT test.
3. Polyglandular auto immune disease, Addison's disease, pernicious anemia, celiac sprue. Note: Investigators are not mandated to test for Celiac disease (also known as Sprue). Subjects suspected of having Celiac disease should be tested for the presence of disease, as part of good medical care, as treatment would differ. Treated, stable Hashimoto's thyroiditis is not exclusionary.
4. Any of the following abnormal laboratory values at screening: total white blood cell count (WBC) outside the range of 1,500-15,000/mm3 (1.5-15.0 x 109/L), neutrophil count (<1500/mm3) (<1.5 X 109 / L), lymphocyte count <500/mm3 (<0.5 X 109 / L), hemoglobin (Hgb) <8.0 g/dL, platelets <100,000/mm3 (<100 x 109/L) 5. History of immunodeficiency disorders, such as HyperIgM syndrome; history of recurrent infections suggestive of immunodeficiency disorders.

6. History of or active coagulation disorder with increased thromboembolic risk; a PTT and PT/ INR below lower limit of normal prior to inclusion.

7. Tuberculosis infection assessed by positive QuantiFERON TB-Gold test (QFT) at screening. Subjects with a positive QFT test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then anti tuberculosis treatment must have been initiated and maintained according to local country guidelines.

8. Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV). A positive HBV surface antigen (HBsAg) test, at screening, excludes a subject. Subjects with a positive HCV antibody test should have HCV RNA levels measured. Subjects with positive (detectable) HCV RNA should be excluded.

9. Positive human immune virus HIV test (ELISA and Western Blot) at screening. 10. Evidence of EBV, CMV, HSV, and/or SARS-CoV-2 infection by viral load above laboratory upper limit of normal or only positive IgM serology in the absence of positive IgG at screening. Rescreening is permitted in persistently asymptomatic or postsymptomatic subjects, but study drug must be able to be administered within 100 days of diagnosis of T1D and viral load must be negative and IgG titers positive.

11. Major dental work (e.g. tooth extractions or dental surgery with access to dental pulp) within 8 days of first dose; febrile illness within 48 hrs of first dose.

12. Use of other investigational drugs or use of immunosuppressive agents at the time of enrollment, or within 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.

13. History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study. Multiple and recurring allergies refer to known allergies to the investigational compound, to immunoglobulin based therapies, or to multiple drug classes. Dust mites, hay fever, and similar environmental allergies are not exclusionary.

14. History of severe hypersensitivity reaction or anaphylaxis to biological agents, e.g. human monoclonal antibody.

15. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.

16. Active serious psychiatric disorders (diagnosed or treated by a psychiatrist), such as eating disorders and psychosis or history thereof.

17. Any complicating medical issues or clinically abnormal laboratory results that may cause an increased safety risk to the subject as judged by the investigator.

18. Ongoing, and up to 2 weeks prior to screening, use of medications that may affect glucose control (e.g, systemic steroids, thiazides, beta blockers). A short course of oral steroids <10 days if medically required is permissible with sponsor notification.

19. History of drug abuse, nicotine or harmful alcohol use within 12 months prior to first dose, or evidence (as determined by the investigators) of such abuse at screening. For example, harmful alcohol use in adults is defined as five or more drinks per day for 5 or more days in the past 30 days. Harmful alcohol use by adolescents (age 13-18 years) is to be determined by the investigator, based on local culture and laws. Harmful cannabinoid use is difficult to define universally and the determination of abuse will be made by the Investigator based on local culture and law.

20. Taking medications prohibited by the protocol 21. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

22. Women of child-bearing potential, defined as all women, who are sexually active, physiologically capable of becoming pregnant (e.g. menstruating), unless they are using highly effective methods of contraception during dosing and for 14 weeks after stopping the investigational drug. Highly effective contraception methods include:

* Total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks prior to first dose. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization in the sexual partner of female study participant (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
* Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
* In case of use of oral contraception, women should be stable on the same pill for a minimum of 3 months prior to first dose.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Augsburg, Germany
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
- Novartis Investigative Site, Ljubljana, Slovenia
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, A Coruña, Galicia
- Novartis Investigative Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 12 investigative sites in 6 countries.
Pre-assignment Details: Enrolment was based on both screening and baseline results. The screening and baseline visit(s) may be conducted over 1 or more visits depending on the subject's body weight and World Health Organization and European Medicines Agency (EMA) recommendations for trial related phlebotomy limits.
Groups:
- CFZ533: CFZ533 30 mg/kg i.v. dose on Day 1. From Day 8 up to Day 358 participants with body weight of ≥30 to <50 kg received 195 mg s.c., and participants with body weight of ≥ 50 kg to ≤125 kg received 300 mg s.c. on a weekly basis.
- Placebo: Placebo i.v. dose on Day 1. From Day 8 up to Day 358 participants with body weight of ≥30 to <50 kg and body weight of ≥ 50 kg to ≤125 kg received matching placebo s.c. on a weekly basis.
Period: Overall Study
Arm/Group | CFZ533 | Placebo
Started | 29 | 15
Completed | 26 | 13
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ533 | Placebo | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (2.81) | 15.5 (3.07) | 15.5 (2.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 19 | 10 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs led to study treatment discontinuation, and SAEs. On-treatment period is defined as from date of first administration of study treatment to 98 days after date of last administration of study treatment (including start and stop date).
Time Frame: Adverse events were reported from first dose of study treatment to 98 days after last dose, up to a maximum duration of approximately 65 weeks.
Population: The safety analysis set included all participants that received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 29 | 15
Participants
  Adverse Events | 28 | 13
  Serious Adverse Events | 4 | 1
  AEs leading to discontinuation of study treatment | 4 | 0

2. Primary Outcome: Normalized Stimulated C-peptide Area Under the Curve (AUC) at Week 52
Description: The mixed meal tolerance test (MMTT) has appropriate sensitivity to detect residual insulin secretion and beta cell function. In the MMTT, following an 8-10 hour overnight fast, a weight-based liquid meal provided as 6 mL/kg (maximum 360 mL) of mixed meal, ingested over 5 min with timed blood samples for glucose and C peptide determination obtained 10 min prior to ingestion (t = -10), at baseline (t = 0), and at 15, 30, 60, 90, and 120 min after consumption of the liquid meal. The time collections for post load samples are based on the start time of the mixed meal.
  Stimulated C-peptide AUC by the standard MMTT, normalized by the duration of measurements, was analyzed with a mixed model repeated measures analysis.
Time Frame: At Week 52, 10 min prior to ingestion, at start of ingestion, and at 15, 30, 60, 90, and 120 min after consumption of the liquid meal.
Population: The full analysis set (FAS) included all participants to whom study treatment has been assigned by randomization.
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: nmol/L
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 29 | 15
nmol/L | 0.42 [0.36 to 0.49] | 0.36 [0.30 to 0.44]
Statistical Analysis 1: Comparison: CFZ533 vs Placebo; Test type: Superiority; p = 0.1817, Mixed model repeated measure analysis — one-sided P-value; Ratio of geometric means CFZ533/placebo = 1.173, 80% CI 2-sided [0.94 to 1.47]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of CFZ533 After Intravenous (IV) Administration
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. Free CFZ533 plasma concentrations were determined using a validated target-based sandwich enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Day 1: Pre-dose and 90 minutes after the start of the IV infusion (duration of the infusion is 30 minutes).
Population: The pharmacokinetic (PK) analysis set included all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any dose of CFZ533 and with no protocol deviations that impact on PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533
Number analyzed (Participants) | 29
ug/mL | 506 (124)

4. Secondary Outcome: Trough Plasma Concentration (Ctrough) of CFZ533
Description: Ctrough is the observed plasma concentration that is just prior to the beginning of, or at the end of a dosing interval. Free CFZ533 plasma concentrations were determined using a validated target-based sandwich ELISA method.
Time Frame: Pre-dose at: Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, Week 56, Week 60, Week 64, Week 68, Week 72.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CFZ533
Number analyzed (Participants) | 29
ug/mL
  Day 1: number analyzed (Participants) | 27
  Day 1 | 0.00 (0.00)
  Week 4: number analyzed (Participants) | 26
  Week 4 | 182 (40.9)
  Week 8: number analyzed (Participants) | 25
  Week 8 | 171 (45.8)
  Week 12: number analyzed (Participants) | 21
  Week 12 | 169 (43.1)
  Week 16: number analyzed (Participants) | 18
  Week 16 | 193 (55.2)
  Week 20: number analyzed (Participants) | 20
  Week 20 | 184 (68.1)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 176 (65.2)
  Week 28: number analyzed (Participants) | 18
  Week 28 | 186 (61.4)
  Week 32: number analyzed (Participants) | 16
  Week 32 | 177 (65.4)
  Week 36: number analyzed (Participants) | 17
  Week 36 | 180 (86.7)
  Week 40: number analyzed (Participants) | 15
  Week 40 | 183 (80.0)
  Week 44: number analyzed (Participants) | 14
  Week 44 | 170 (88.7)
  Week 48: number analyzed (Participants) | 15
  Week 48 | 205 (101)
  Week 52 | 155 (111)
  Week 56: number analyzed (Participants) | 26
  Week 56 | 72.6 (53.3)
  Week 60: number analyzed (Participants) | 25
  Week 60 | 30.9 (24.9)
  Week 64: number analyzed (Participants) | 26
  Week 64 | 9.23 (11.7)
  Week 68: number analyzed (Participants) | 25
  Week 68 | 1.86 (3.15)
  Week 72: number analyzed (Participants) | 26
  Week 72 | 0.221 (0.499)

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of CFZ533 After IV Administration
Description: Tmax is the time to reach maximum (peak) drug concentration after single-dose administration (time). Free CFZ533 plasma concentrations were determined using a validated target-based sandwich ELISA method. Theoretical sampling time points were used to report Tmax.
Time Frame: Day 1: Pre-dose and 90 minutes after the start of the IV infusion (duration of the infusion is 30 minutes).
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | CFZ533
Number analyzed (Participants) | 29
hours | 1.5 [1.5 to 1.5]

6. Secondary Outcome: Number of Participants With Full or Partial Remission
Description: Full remission is defined by HbA1c ≤ 6.5% (48 mmol/mol) and no exogenous insulin use at Week 52.
  Partial remission 1 is defined by Insulin Dose Adjusted HbA1c (IDAA1c) ≤ 9.0 at Week 52.
  Partial remission 2 is defined by HbA1c < 7.0% (53 mmol/mol) and total daily insulin dose <0.5 units per kg per day at Week 52.
  Two different criteria for partial remission were considered, and patients were assessed separately according to each criterion.
Time Frame: Week 52
Population: The full analysis set (FAS) included all participants to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 29 | 15
Participants
  Full remission* | 0 | 0
  Partial remission 1 | 20 | 10
  Partial remission 2 | 15 | 6

7. Secondary Outcome: Normalized Stimulated C-peptide Area Under the Curve (AUC) at Week 72
Description: as for outcome 2
Time Frame: At Week 72, 10 min prior to ingestion, at start of ingestion, and at 15, 30, 60, 90, and 120 min after consumption of the liquid meal.
Population: The full analysis set (FAS) included all participants to whom study treatment has been assigned by randomization.
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: nmol/L
Arm/Group | CFZ533 | Placebo
Number analyzed (Participants) | 29 | 15
nmol/L | 0.40 [0.34 to 0.47] | 0.32 [0.26 to 0.39]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 72 weeks.
Groups:
- Total: Total
Arm/Group | CFZ533 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15 | 0/44
Serious Adverse Events (participants affected / at risk) | 6/29 | 1/15 | 7/44
Other Adverse Events (participants affected / at risk) | 27/29 | 14/15 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 (N=29) | Placebo (N=15) | Total (N=44)
Pyrexia (General disorders) | 1 | 0 | 1
Large intestine infection (Infections and infestations) | 1 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Tonic clonic movements (Nervous system disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 (N=29) | Placebo (N=15) | Total (N=44)
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 4
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 2 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Asthenia (General disorders) | 1 | 1 | 2
Injection site reaction (General disorders) | 7 | 3 | 10
Malaise (General disorders) | 0 | 1 | 1
Medical device pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 5 | 3 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 1 | 2
COVID-19 (Infections and infestations) | 7 | 2 | 9
Chronic active Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 2 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 3 | 3 | 6
Nasopharyngitis (Infections and infestations) | 13 | 5 | 18
Otitis externa (Infections and infestations) | 1 | 1 | 2
Parvovirus B19 infection (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 2
Pharyngotonsillitis (Infections and infestations) | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Rhinitis (Infections and infestations) | 2 | 2 | 4
Sinusitis (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 2 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 3 | 3
Tooth abscess (Infections and infestations) | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 7
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Viral infection (Infections and infestations) | 2 | 0 | 2
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 3
Lipids increased (Investigations) | 1 | 1 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1
Serology positive (Investigations) | 2 | 0 | 2
Urine analysis abnormal (Investigations) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 19 | 8 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Headache (Nervous system disorders) | 7 | 2 | 9
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04129528/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04129528/SAP_001.pdf